CLINICAL TRIAL: NCT01673074
Title: A Phase 1 Trial of Photodynamic Therapy With HPPH in Patients With Pleural Malignancy
Brief Title: HPPH and PDT for Pleural Malignancy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: UPCC 02507
Record Dates: First submitted 2012-08-20; First posted 2012-08-27 (Estimated); Last update posted 2020-04-08 (Actual); Status verified 2020-04

CONDITIONS: Pleural Malignancy
MeSH Terms: interventions — Ultraviolet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: (PDT) Photodynamic therapy — photosensitizer

SUMMARY:
The primary objective of the study is to determine the maximally tolerated photodynamic therapy (PDT) dose and drug-light interval of PDT using light and HPPH in patients with pleural malignancy who have undergone a maximal resection.

DETAILED DESCRIPTION:
Photodynamic therapy (PDT) is an experimental treatment that uses a drug called a photosensitizer or photosensitizing agent and light to kill cells. When photosensitizers are exposed to a specific wavelength of light, they produce a form of oxygen that kills hearby cells. The appeal o PDT in oncology has been that the photosensitizer is retained in tumor tissue for longer periods of time compared to normal tissues. This reported differential of photosensitizer retention in tumor compared to normal tissues provides the potential for an enhanced therapeutic index minimizing normal tissue toxicity has prompted an interest in studying PDT as a cancer treatment and is a proposed treatment for a variety of malignancies and pre-malignant conditions. The proposed study is a Phase I trial of photodynamic therapy (PDT) for the treatment of patients with pleural malignancies. To participate patients must be 18 years of age or older, must have a histological diagnosis of pleural malignancy, must have disease limited to the hemithorax (one side of the chest), must be medically suitable for resection, and must have a ECOG performance status of 0-2. Patients who have received prior surgery, gene therapy, or combination chemotherapy will also be permitted if it has been at least 30 days since the last treatment. Patients will be given HPPH, by intravenous injection prior to surgery. HPPH is a chlorine based photosensitizer used along with PDT to prevent recurrence of tumors following surgical removal. After successful tumor removal light from a tunable dye laser or diode laser will be administered. The starting dose of PDT will ve administered 24 or 48 hours prior to surgical resection. Red light will be used to illuminate the entire thoracic cavity. If adequate removal of the tumor cannot be performed , the patient will not be eligible to receive light therapy. In parallel laboratory studies, biopsies of tumor and normal tissues will be taken from the resection specimens. Uptake of HPPH will be measured in tumor and normal tissues and tumor to normal tissue ratios of HPPH will be determined. Assessment of molecular signaling including EGFR, Akt, and MAPK will be made in tumor prior to and after light delivery. Patients will simultaneously be enrolled on a companion protocol in which the 2-nitroimidazole, EF5 will be administered to determine tumor oxygen concentration. Finally, non-invasive measurements of optical properties, tissue oxygenation, photosensitizer uptake, and blood flow will be made intraoperatively. After hospital discharge patients will be seen routinely in outpatient Thoracic Surgery and Radiation Oncology Department clinics. These follow visits will occur one month., two months later and every three months of the first 24 months to assess treatment related toxicities. A history and physical examination, laboratory and a CT or MRI of the chest will be performed every 3 months. A follow-up chest x-ray will be obtained as clinically indicated. An assessment of toxicity will be made at each follow-up visit. After 24 months, follow-up should be scheduled as clinically indicated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a histologic diagnosis of a pleural malignancy who in the opinion of the attending thoracic surgeon can be resected to a maximal thickness of < 0.5cm. Patients must have disease limited to the hemithorax. Patients whonhave received prior surgery, gene therapy, or combination chemotherapy will be permitted if it has been at least 30 days since the last treatment. Patients may receive post-operative chemotherapy or radiation therapy after completion of surgery and PDT if these treatments are clinically indicated.
* ECOG performance status of 0-2.
* Medical suitability for resection.
* 18 years of age or older.
* Patients must sign a document that indicates that they are aware of the investigative nature of the treatment of this protocol and the potential benefits and risks. Patients unwilling to sign informed consent are excluded from the study.
* All cell types of pleural malignancy will be included.

Exclusion Criteria:

* Patients with active co-existing malignancy are excluded.
* Pregnant or lactating patients.
* Patients who have a history of HIV disease.
* Patients who have a white count less than 2500 per cubic mm or platelets less than 100,000/cubic mm.
* Serum creatinine equal or greater than 2.5 mg/deciliter. Patients who have severe liver disease including cirrhosis, Grade III-IV elevations in liver function studies, or bilirubin in excess of 1.5 mg/deciliter.
* Patients with porphyria or hypersensitivity to porphyrin or porphyrin-like compounds.
* Patients who have received prior mantle radiation.
* Patients who have received Alimta<8 weeks prior to surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2007-11; Primary Completion 2013-12 (Actual); Study Completion 2014-10-08 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Keith Cengel, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States